CLINICAL TRIAL: NCT06447194
Title: Effect of Local Injectable Ropivacaine, Epinephrine, Clonidine, and Ketorolac (RECK) Anesthetic Cocktail on Postoperative Pain in Posterior Spinal Fusion
Brief Title: Effect of RECK in Posterior Spinal Fusion
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was not feasible due to logistical and implementation challenges. No participants were enrolled and the study will not proceed further.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Steven Ludwig, Professor, Department of Orthopaedics, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00109268
Record Dates: First submitted 2024-05-14; First posted 2024-06-07 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Degenerative Lumbar Spinal Stenosis; Degenerative Disc Disease; Degenerative Spondylolisthesis; Degenerative Disease
Keywords: Spine Surgery; Lumbar Fusion; Pain Control; Opioid Utilization; Local Anesthesia; RECK; R.E.C.K.; Ropivacaine; Epinephrine; Clonidine; Ketorolac; Randomized Controlled Trial
MeSH Terms: conditions — Intervertebral Disc Degeneration; Agnosia | interventions — Ropivacaine; Epinephrine; Clonidine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded by investigational drug service
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (RECK) (Experimental): The arm of patients who will be administered "RECK" local anesthesia cocktail:
  Ropivacaine 0.125g Clonidine 80 mcg Epinephrine 0.5 mg Ketorolac 30 mg In sterile water 73 mL (total volume of compound is 100 mL)
  Given through paraspinal muscle injection once intraoperatively.
  Interventions: Drug: Ropivacaine, Epinephrine, Clonidine, and Ketorolac Injection Cocktail
- Control Group (Placebo) (Placebo Comparator): The arm of patients who will be administered a placebo injection:
  100 mL Normal Saline
  Given through paraspinal muscle injection once intraoperatively.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ropivacaine, Epinephrine, Clonidine, and Ketorolac Injection Cocktail — Please refer to description for interventional group.
  Other Names: RECK
  Arms: Intervention (RECK)
Other: Placebo — 100mL paraspinal normal saline injection intraoperatively, once.
  Arms: Control Group (Placebo)

SUMMARY:
"RECK" is a combination of local anesthesia medications, used for the purpose of pain control. RECK is an acronym which stands for Ropivacaine, Epinephrine, Clonidine, and Ketorolac. The purpose of this study is to investigate the effect of RECK local injectable anesthetic in the setting of posterior spinal fusion. Our specific aims are the following.

Primary aim: to investigate the effect of RECK local injectable anesthetic on postoperative VAS pain scores.

Secondary aims: to investigate of effect of RECK injection on postoperative opioid consumption and hospital length of stay.

Hypothesis: RECK injection will significantly decrease postoperative VAS pain score, opioid consumption, and hospital length of stay compared to placebo controls.

DETAILED DESCRIPTION:
Patients will be randomized into two groups. Intraoperatively, they will be given either 1) a 50 mL RECK (ropivacaine, epinephrine, clonidine, and ketorolac) cocktail containing 123 mg ropivacaine, 0.25 mg epinephrine, 0.04 mg clonidine, and 15 mg ketorolac into the paraspinal musculature and subdermal space surrounding the operative site once the fascia is closed (intervention group), or 2) a 50 mL injection of saline (control group). RECK is used for pain control and will be administered by fellowship-trained orthopaedic spine surgeons. All patients will have a patient-controlled analgesia pump initiated shortly after surgery, with routine postoperative care and observation from nurses, pain management, and orthopedic surgeons and residents.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-88 years old
* Undergoing spinal fusion at 1-3 lumbar levels via a posterior approach.

Exclusion Criteria:

* Revision surgeries
* Surgeries indicated for trauma, tumor, or infection
* Preoperative history of moderate to severe hepatic, renal, cardiac, or psychiatric illness
* Known hypersensitivity to any of the RECK components

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative VAS Pain Scores | 2, 4, and 6 hours immediately postoperatively, then repeating once daily through hospital admission (an average of 4 days)
  Primary aim: to investigate the effect of RECK local injectable anesthetic on postoperative VAS pain scores.
  VAS (Visual Analogue Scale) measures pain intensity. The VAS is a 10cm line with two end points representing 0 ("No pain") and 10 ("Pain as bad as it could be"). The patient is asked to rate their pain by placing a marker on the line. A lower score (thus closer to "no pain") is a better outcome.

SECONDARY OUTCOMES:
Opioid Utilization | Postoperatively day 1, then repeating once daily through hospital admission (an average of 4 days)
  Secondary aims: to investigate of effect of RECK injection on postoperative opioid consumption.
Hospital Length of Stay | Up to 2 weeks (an average of 4 days)
  Secondary aims: to investigate of effect of RECK injection on hospital length of stay.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No